CLINICAL TRIAL: NCT06714344
Title: A Prospective Open Randomised Trial to Test the Efficacy of an Assisted Therapy
Brief Title: Efficacy of an Assisted Therapy Optimizing Module to Improve Physician Adherence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: AIT Austrian Institute of Technology GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AMPEL
Record Dates: First submitted 2024-11-13; First posted 2024-12-03 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMPEL group (Experimental): Network physicians participating in the study are randomly assigned to the AMPEL group (access to the module).
  Interventions: Device: KITGuideMe: W61-MD41-AIT, version 1.0.0
- non-AMPEL group (No Intervention): The non-AMPEL group (no access to the module) using a permuted block randomization scheme to ensure that there are the same number of patients in each study arm.

INTERVENTIONS:
Device: KITGuideMe: W61-MD41-AIT, version 1.0.0 — We are planning to conduct a prospective, 1:1 randomized study within the HM program.
  Randomization occurs at the level of network physicians. Network physicians participating in the study are randomly assigned to either the AMPEL group (access to the module) or the non-AMPEL group (no access to the module) using a permuted block randomization scheme to ensure that there are the same number of patients in each study arm. Logical checks within the module ensure that once a network physician is assigned to an arm, he or she remains in that arm for the remainder of the stud
  Arms: AMPEL group

SUMMARY:
Heart failure patients within the HM programme

DETAILED DESCRIPTION:
A prospective, randomized, multi-sectoral multi-centre study with parallel group design.

Application of guideline-directed medical therapy (GDMT) improves quality of life and decreases hospitalization for heart failure and mortality.

GDMT is in general underused. This also applies to patients who are cared for in the integrative, telemedicine-supported disease management program Herzmobil Tirol (HMT). The Assisted Therapy Optimizing Module has been designed to actively assist network physicians in adhering to and improving guideline-based medical therapy.

ELIGIBILITY:
Inclusion Criteria:

AMPEL, CIP, Version: 1.2 Date: 27.03.2024

1. Written, signed and dated informed consent for inclusion in the HM programme
2. Male and female patients over 18 years of age.
3. Hospitalised for decompensated heart failure requiring intravenous diuretics
4. Need for iv diuresis in nonhospital setting because of impending hospitalization for cardiac decompensation

Exclusion Criteria:

1. Multimorbidity (Charlson Comorbidity Index > 6)
2. Dementia
3. Lack of willingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female patients
Enrollment: 234 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoints | 09/2027
  The therapy optimization module improves guideline compliance within the framework of the Herzmobil care program individually optimized number and dose of GDMT 90 days after randomization based on the GDMT score. individually optimized number and dose of GDMT 90 days after randomization based on the GDMT score.

SECONDARY OUTCOMES:
Secondary Endpoints | 09/2027
  Increased guideline-based therapy will reduce mortality and rehospitalization rates.
  admissions vs. non-cardiovascular admissions) after 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Medical University of Graz, University Hospital for Internal Medicine (Cardiology), Graz, Styria
  - Medical University of Innsbruck, University Hospital for Internal Medicine III (Cardiology and Angiology), Innsbruck, Tyrol